CLINICAL TRIAL: NCT06062433
Title: Assessment of Feasibility and Effectiveness of Remote Asthma Management Via an Integrated Artificial Intelligence-assisted Clinical Decision Support System With Mobile Device Compared With Usual Asthma Care in Pediatric Participants With Asthma Aged 6-17 Years: A Parallel Group, Non-blinded, Dual-site, 2-arm, Pragmatic Randomized Clinical Trial
Brief Title: A Study of Remote Asthma Management Using an Integrated Artificial Intelligence-assisted EHR Dashboard and Mobile Device Compared With Usual Asthma Care to Treat 6-17 Year Old Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Young Juhn, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-001438
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Pediatric Asthma Intervention Group (Experimental): Along with clinical standard of care for asthma, subjects will have Asthma-Guidance and Prediction System (A-GPS) with AsthmaTuner (AT) integrated into care.
  Interventions: Device: AsthmaTuner; Other: Asthma-Guidance and Prediction System
- Pediatric Asthma Control Group (No Intervention): Subjects will receive clinical standard of care for asthma.
- Clinician Control Group (No Intervention): Clinicians will provide clinical standard of care for pediatric asthma patients.
- Clinician Intervention Group (Experimental): Clinicians will integrate Asthma-Guidance and Prediction System (A-GPS) with AsthmaTuner (AT) into clinical standard of care for asthma.
  Interventions: Device: AsthmaTuner; Other: Asthma-Guidance and Prediction System
- Asthma Care Coordinator Control Group (No Intervention): Asthma Care Coordinators will provide clinical standard of care for pediatric asthma patients.
- Asthma Care Coordinator Intervention Group (Experimental): Asthma Care Coordinators will integrate Asthma-Guidance and Prediction System (A-GPS) with AsthmaTuner (AT) into clinical standard of care for asthma.
  Interventions: Device: AsthmaTuner; Other: Asthma-Guidance and Prediction System

INTERVENTIONS:
Device: AsthmaTuner — Phone application and spirometer for self-management of asthma
  Other Names: AT
  Arms: Asthma Care Coordinator Intervention Group; Clinician Intervention Group; Pediatric Asthma Intervention Group
Other: Asthma-Guidance and Prediction System — Artificial Intelligence (AI)-assisted clinical decision support system which extracts pertinent patient data related to asthma management from electronic health record
  Other Names: A-GPS
  Arms: Asthma Care Coordinator Intervention Group; Clinician Intervention Group; Pediatric Asthma Intervention Group

SUMMARY:
The main purpose of this study is to look at whether clinicians and their patients with asthma can satisfactorily perform remote asthma management at home (not visiting clinic) by using an artificial intelligence tool called Asthma-Guidance and Prediction System combined with a home monitoring device called AsthmaTuner.

ELIGIBILITY:
Inclusion Criteria:

Clinician participants are eligible to be included in the study only if all of the following criteria apply:

* Employed as consultant or nurse practitioner at study sites.
* Able to provide written consent.
* Are willing to follow recommendations to schedule/see participant and their caregiver for regular asthma follow-up care every 3-6 months.

All asthma care coordinators who are involved in the usual care of pediatric participants will also be recruited for inclusion in the study.

Pediatric participants are eligible to be included in the study only if all of the following criteria apply:

* Ages 6-17 years old with diagnosis of asthma.
* Have a caregiver who is willing to participate alongside pediatric participant and to have regular asthma follow-up care every 3-6 months.
* Adolescent participants ages 13-17 years and their caregivers are able to give written informed consent; or child participants ages 7-12 years are able to provide assent and their caregivers are able to give written informed consent (subjects who are 6 years old will be waived).
* Both participant and caregiver are able to read and write in English.
* Receive pediatric primary care at study sites from participating study clinician.
* Access for caregiver and/or adolescent participants to an Android or iPhone with Wi-Fi access and availability for at least monthly use.
* Active asthma defined by at least one clinic visit with a diagnosis of asthma per EHR or on active asthma control or rescue medication in the past 12 months. Priority will be given to those with persistent asthma on inhaled corticosteroids therapy or those with poorly controlled asthma defined by any of the following criteria in the past 12 months, except item v (past 2-week period); i. Asthma Control Test for adolescents ≥ 12 years or Childhood Asthma Control Test for children < 12 years (score< 20); ii. ED visit for asthma; or iii. Hospitalization for asthma; or iv. Unscheduled outpatient visit for asthma requiring oral corticosteroid use; or v. Asthma symptoms at the screening interview, including 1) more than 2 days per week shortness of breath, wheezing, chest tightness, or 2) more than 1 night awakening due to asthma in the past 2-week period.
* Participant had their latest asthma follow-up visit more than 3 months prior to the screening date of the study.

Exclusion Criteria:

Pediatric participants who do not meet the eligibility criteria described above will be excluded and those will be excluded from the study if any of the following criteria apply:

* Major medical problems prohibiting study participation and inability to perform study procedures (including spirometry); suspected symptoms of exercise-induced laryngeal obstruction (EILO), tracheobronchial foreign body at or about the incidence date of asthma, wheezing occurring only in response to anesthesia or medications, bullous emphysema or pulmonary fibrosis on chest radiograph, PiZZ alpha1-antitrypsin, cystic fibrosis, or other major chest disease such as severe kyphoscoliosis or bronchiectasis.
* Pediatric participant pregnancy.
* Hyposensitization therapy for > 3 months prior to study enrollment.
* Participation in any other interventional studies for asthma within 1 month prior to study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Change in satisfaction of asthma care | Baseline, 6 months
  Measured by single question to assess satisfaction about asthma care using a Likert scale where 1=strongly disagree and 5=strongly agree. Higher score indicates greater satisfaction.

SECONDARY OUTCOMES:
Time allocated to asthma visits | 6 months
  Total time allocated to asthma visits which includes time spent with pediatric participant, EHR review, and completion of timed clinical task.
Number of on-site visits | 6 months
  Total number of on-site visits for related asthma care
Frequency of poorly controlled asthma | Baseline, 6 months
  Number of subjects to have poorly controlled asthma defined as Asthma Control Test or Childhood Asthma Control Test score less than 20.

CONTACTS AND LOCATIONS:
Overall Officials: Young Juhn, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Myers L, Brereton TA, Overgaard S, Greenwood JD, Zheng L, Ohde JW, Spiten M, Kathy Ihrke RN, Lang K, Peterson K, Hawley S, Beenken M, Malik M, Bublitz J, Galloway T, Wilkes Q, Shrader D, Mercado L, Park M, Arteta M, Hartz M, Fladager-Muth J, Quam M, Perrigo T, Loufek T, Khurana A, Kshatriya BSA, Sharma D, Le-Rademacher J, Wi CI, Nordlund B, Juhn Y. Pediatric asthma management via integration of a remote spirometry device into an EHR-based artificial intelligence-powered clinical decision support system: A feasibility pragmatic clinical trial. Contemp Clin Trials. 2025 Dec 24;161:108209. doi: 10.1016/j.cct.2025.108209. Online ahead of print. PMID 41453519
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials